CLINICAL TRIAL: NCT00971503
Title: Método Para Regenerar el páncreas Con localización in Vivo de médula ósea Total Autologa en Pacientes diabéticos Tipo 1. Estudio Fase IIB.
Brief Title: Safety and Efficacy of Arterial Delivery of Autologous Bone Marrow Cells in the Treatment of Insulin-Dependent Diabetes
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator moved to Chile from Argentina
Sponsor: University of Moron (Other)
Responsible Party: BMG Biotech
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CM 02
Record Dates: First submitted 2009-09-01; First posted 2009-09-03 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Diabetes type 1; Adult Stem cells; Local injection; Catheter delivery; Bone marrow
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saline injection (Sham Comparator)
  Interventions: Other: Saline injection
- Autologous bone marrow implantation (Experimental)
  Interventions: Procedure: autologous bone marrow implantation

INTERVENTIONS:
Procedure: autologous bone marrow implantation — Filgrastim treatment before bone marrow aspiration that will then be implanted via pancreatic artery
  Arms: Autologous bone marrow implantation
Other: Saline injection — Injection of saline solution for 5 days
  Arms: saline injection

SUMMARY:
Diabetes mellitus is a long-term multi-organ disease with severe implications that constitute a major health problem worldwide. Type 1 diabetes is an autoimmune disorder in which the body's own immune system attacks and destroys the cells that make insulin. Exogenous administration of insulin is the primary method of controlling type 1 diabetes by regulating blood glucose levels, but this treatment does not reverse nor prevent disease progression.

Our hypothesis is that when implanting stimulated total bone marrow by arterial injection directly into the pancreas, we will achieve functional recovery of insulin-producing cells. This study will include patients with chronic type 1 diabetes and absence of lesions in target organs. We will follow the evolution of patients receiving autologous total bone marrow implantation by selective catheterization and compare to a non-treatment control group. All subjects will continue to use insulin therapy as needed to maintain the best possible glucose control.

The objective is to achieve a significant increase in C-peptide levels indicating a regeneration of the beta islet cells with a decrease in exogenous insulin usage in at least 70% of the patients.

This study is a follow-up to our initial study in which 22 patients received autologous total bone marrow. The initial study was 100% safe but additional studies like the one described above are needed to show efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Between 18-30 years of age, diagnosed with diabetes mellitus Type 1 (insulin-dependent).
* Negative antibody titers for GAD and anti-islet.
* Measurements of serum C-peptide below normal values.
* BMI 20-25, men, 19-24, women

Exclusion Criteria:

* Diabetes type 2, gestational diabetes, and other types of secondary diabetes.
* Patients with acute metabolic complications of diabetes such as ketoacidosis at least within the last 6 months.
* Abdominal perimeter >102 cm in men; >88cm in women
* Fasting glycemia >100 mg/dl, triglycerides >150 mg/dl, HDL < 40 mg/dl.
* Blood pressure: SBP >135 mmHg and DBP >85 mmHg at the time of randomization
* Patients with BMI > 25 for men and >24 for women.
* Patients weighing < 40 kg.
* Patients with abnormal ECG indicative of acute or chronic ischemia or acute/chronic necrosis.
* Patients with anemias of any origin.
* Patients undergoing antibiotic treatment for acute infection.
* Patients with any blood abnormality.
* Patients with history of moderate to severe pancreatitis.
* A female subject who is breast-feeding, pregnant, intends to become pregnant or refuses to use a contraceptive method during the course of the study.
* Patients allergic to iodine or filgrastim.
* Patients using medications that could affect this study.
* Patients with serious mental conditions.
* Patients who have undergone a previous stem cell treatment.
* Patients who do not accept and sign the informed consent.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Significant increase in C-peptide levels after transplant in 70% of the patient. | 1 month, 3 months, 6 months, 12 months, 18 months, 24 months

SECONDARY OUTCOMES:
Reduction by 50% of the insulin requirement after the transplant in 70% of the patients. | Two years
Normalization of the hemoglobin A1C after transplant in 70% of the patients. Normalization of blood glucose levels. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro D. Mesples, MD, Principal Investigator — University of Morón, School of Medicine
Locations (1):
- School of Medicine, Pontificia Universidad Catolica de Chile, Santiago, Santiago de Chile, Chile